CLINICAL TRIAL: NCT04940702
Title: Effectiveness of Focal Vibration and Blood Flow Restriction Within a Multicomponent Exercise Programme for Non-dependent and Sedentary Elderly People. Effects on Biochemical Markers and Functional Tests. Pilot Study.
Brief Title: Effectiveness of Focal Vibration and Blood Flow Restriction Within a Multicomponent Exercise Programme.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER202107
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-06

CONDITIONS: Sarcopenia; Occlusion; Vibration; Exposure; Old Age; Atrophy; Exercise Addiction
MeSH Terms: conditions — Sarcopenia; Bites and Stings; Atrophy | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focal Vibration Group (Experimental): Training with Focal Vibration on rectus anterior, vastus medialis and vastus lateralis muscles with an intensity of 120 Hz and an amplitude of 1.2 mm. Time of training 20-25 min.
  the training is the same as the contol group with the difference of FV addiction.
  Interventions: Other: Focal Vibration
- Blood Flow Restriction Group (Active Comparator): Training with Blood Flow Restriction a pressure cuff occludes in the proximal part of the lower limb. Time of training 20-25 min.
  the training is the same as the contol group with the difference of BFR addiction.
  Interventions: Other: Blood Flow Restriction
- Training Group (Active Comparator): Traditional training. 3 times a week
  1. Warm-up:
  2. Main work:
     1. Aerobic training
     2. Strength training
     3. Balance and coordination training
  3. Return to calm
  Interventions: Other: Traditional Training

INTERVENTIONS:
Other: Focal Vibration — Training with Focal Vibration on rectus anterior, vastus medialis and vastus lateralis muscles with an intensity of 120 Hz and an amplitude of 1.2 mm. Time of training 20-25 min.
  The exercise is the same than traditional training group.
  Arms: Focal Vibration Group
Other: Blood Flow Restriction — Training with Blood Flow Restriction, the restriction is in the proximal part of the lower limb. The exercise is the same than traditional training group.
  Arms: Blood Flow Restriction Group
Other: Traditional Training — Warm up, aerobic training, stenght training, balance and coordination training and return to calm
  Arms: Training Group

SUMMARY:
Sarcopenia can occur or increase due to sedentary lifestyles, physical inactivity or chronic endocrine and inflammatory disorders, this pathology is much more frequent in older people due to the added risk factors and the fact that the physiological ageing process generates a pro-inflammatory situation and an alteration in the synthesis of hormones and myokines, it has been observed that the loss of strength causes functional deterioration and a significant increase in the person's dependence, reduces their functional status and quality of life, and may increase the risk of falls, thereby increasing mortality.

Blood flow restriction (BRR) and focal vibration (FV), which aim to achieve muscular hypertrophy without the need to use high loads or intensities, VF or BFR brings improvements to elderly people with sarcopnoea.

The hipotesis of this study is the addition of BFR or VF techniques to training results in greater improvements in circulating myokine concentrations and functional tests than not adding it.

This study has the objective to determinate whether biochemical markers in serology are able to correlate with improvements in strength, also to study whether the plasma levels of apelin, myomyostatin and lL6 are modified with entraining, to determine whether plasma levels of apelin, myomyostatin and lL6 are further increased by training associated with VF and/or BFR and evaluate the effectiveness of different interventions in improving functional tests.

The methodology of the study is a single-blind, randomised, clinical trial will be conducted. The study population is people over 65 years of age, sedentary, with functional independence and with a state of health that allows them to carry out physical activity. The study is planned as a pilot study and will consist of 30 subjects distributed in: 10 people in the control group (CG), 10 in the experimental vibration group (GE-V) and 10 in the experimental group with restriction (GE-R).

The variables to be measured are anthropometric variables, biochemical markers, variables of neuromuscular function, information about fragility and independence, an functionality.

The intervention will be a training in the control group, the FV and BFR groups will be 3 times a week, with a warm-up, a main block with aerobic work, strength work and training and coordination work, and finally a return to calm, in the experimental groups the strength work will be carried out with these instruments.

DETAILED DESCRIPTION:
The normal ageing process is characterised by a progressive loss of muscle mass and function, this physiological process is known as sarcopenia. As a result of this loss of muscle mass and reduced efficiency of muscle enzymes, a reduction in overall strength and isometric strength in particular is observed. Secondarily, sarcopenia can occur or increase due to sedentary lifestyles, physical inactivity or chronic endocrine and inflammatory disorders. This pathology is much more frequent in older people due to the added risk factors and the fact that the physiological ageing process generates a pro-inflammatory situation and an alteration in the synthesis of hormones and myokines.

Different epidemiological studies show that maximum isometric voluntary contraction is usually maintained up to 45 years of age but its effectiveness decreases with age (25% at 65 years of age and 35% at 70 years of age). When this loss of strength or muscle mass occurs in the elderly with a baseline state of greater frailty or dependence, the clinical importance of this reduction in strength and muscle mass is much more relevant. It has been observed that the loss of strength causes functional deterioration and a significant increase in the person's dependence, reduces their functional status and quality of life, and may increase the risk of falls, thereby increasing mortality. For example, when hospital admissions occur, muscle mass decreases rapidly and in patients with femur fractures and sarcopenia it has been observed that between fracture and hospital discharge (10 days) the Barthel index decreases between 54.7% and 59.5%.

There does not seem to be a clear consensus on the diagnostic criteria for sarcopenia. Anthropometric parameters such as Skeletal Muscle Mass Index (SMMI) (≤8.87 for men and ≤6.42 for women), functional tests such as gait speed (≤0.8 metres/second) or grip strength (<30 or 20 kg for men and women respectively) are some of the most commonly used parameters in the literature for both diagnosis and monitoring of sarcopenia.

To a lesser extent, muscle cross-sectional area or contractile properties of muscle tissue could also be related to this loss of strength. More recently, and with the aim of confirming both the diagnosis and monitoring of sarcopenia, different biochemical markers have been proposed .

Regarding the treatment of sarcopenia, although there are pharmacological approaches to increase or maintain strength and muscle mass, physical activity and nutrition remain the "gold standard". Decreased physical activity level is a major aggravator of sarcopenia and sedentary lifestyles have been shown to result in accelerated loss of muscle mass, strength and functional capacity. Therefore, the American College of Sports Medicine, as well as recent research, shows that strength work at moderate to high load intensity can stimulate bone and muscle metabolism and improve overall strength, gait speed, quality of life, and reduce the risk of falls and cognitive impairment.

Despite the benefit of training at these loads, not all older people are able to perform these activities. This is due to their bone or general fragility, as well as the mechanical stress that this type of exercise produces in their joints or sedentary lifestyles. For these reasons, different types of training have emerged in rehabilitation medicine, such as blood flow restriction (BRR) and focal vibration (FV), which aim to achieve muscular hypertrophy without the need to use high loads or intensities.

BFR is training in which exercise is performed with minimal or no resistance while a pressure cuff occludes the proximal part of the limb. This situation results in partial restriction of arterial flow and more significantly venous flow in the muscles. Given the light or no load applied and the muscle hypertrophy obtained, the BFR is an effective training tool. The BFR avoids the high levels of joint stress and cardiovascular risks associated with high-load training. In the field of sports, the effects of BFR have been extensively studied and, although to a lesser extent, benefits have also been studied in the improvement of physical fitness and rehabilitation of older people.

The use of general or focused vibration is not new in the rehabilitation or de-training field. Vibration is intended to stimulate neuromuscular uses to produce involuntary and additional contractions of muscle tissue, indirectly causing an increase in strength or muscle mass, improving the prevention of falls. This type of equipment has been used both in athletes and in patients with chronic diseases or in intensive care units. There are studies that use vibration in critically ill patients as a safe and feasible intervention for dependent patients. One of the advantages of FV is that it can be used for both unloading and loading, which allows a wide range of adaptation to each patient.

Despite the observed efficacy of VF and BFR, evidence is scarce and no studies have been found to demonstrate that these devices improve the benefits of a multicomponent programme in elderly people with sarcopenia. Noeither have data been located on whether changes in biochemical markers and viscoelastic parameters are sufficiently accurate in observing increases in strength and improvements in muscle tissue.

For all these reasons, the present investigation for objectify to determine whether the use of VF or BFR brings improvements to elderly people with sarcopnoea. As well as, if the biochemical and viscoelastic markers can objectify the improvements obtained by means of the multicomponent exercise (with and without the use of BFR and VF).

The hipotesis of this study is the addition of BFR or VF techniques to training results in greater improvements in circulating myokine concentrations and functional tests than not adding it.

This study has the objective to determinate whether biochemical markers in serology are able to correlate with improvements in strength, also to study whether the plasma levels of apelin, myomyostatin and lL6 are modified with entraining, to determine whether plasma levels of apelin, myomyostatin and lL6 are further increased by training associated with VF and/or BFR and evaluate the effectiveness of different interventions in improving functional tests.

The methodology of the study is a single-blind, randomised, clinical trial will be conducted. Pilot study pre and post intervention with control group. Which will follow the CONSORT guide for the implementation of this study and the TIDier guide for the implementation of the intervention.

The study population is people over 65 years of age, sedentary, with functional independence and with a state of health that allows them to carry out physical activity. The study is planned as a pilot study and will consist of 30 subjects distributed in: 10 people in the control group (CG), 10 in the experimental vibration group (GE-V) and 10 in the experimental group with restriction (GE-R).

The variables to be measured are anthropometric variables such as height, sex, age, lower limb dominance and bioimpedance, we will also measure biochemical markers: a complete blood count will assess the levels of: Apelin (primary endpoint), myostatin, IL6, plasma proteins, uric acid and creatinine. Information about physical activity via PASE scale, variables of neuromuscular function, with Tensiomyography: Contraction time (Tc), and radial displacement (Dm), Myotonometry: Stiffness, Surface electromyography: %RMS, all of this in muscles Rectus femoris, vastus lateralis, vastus medialis, lateral gastrocnemius and tibialis anterior. Manual dynamometry: Peak force (Kg). Movements: Knee and hip flexion and extension, plantar flexion and dorsal flexion of the ankle, grip strength (Handgrip), stabilometry and ecography to measure the muscle cross-section.

Information about fragility and independence, with Barthel index, FRAIL scale, Falls Efficacy Scale I (FES-I), SARC-F. Information on functionality with Short Physical Performance Battery (SPPB), velocity in 4 meters walking, Timed get up and go (TUG).

The intervention in the control group, will be a training 3 times a week with, warm up,articular and functional exercises with one's own body weight, principal work: Aerobic training 20 minutes waking then strenght training 25 minutes, i.Sets: start with 1 set to consolidate the technique, and progress to 3 sets.

ii.Repetitions: start with 10-15 repetitions (at lower intensity) and progress to 8-12 repetitions.

iii.Intensity: start with a lower intensity (even 20-30%1RM) and progress to 70-80%1RM.

iv.Rest: Breaks between sets of 3-5 minutes should be taken to avoid muscle fatigue.

v.Exercises: Leg press on machine Balance and co-ordination training during 5-10 minutes finally return to calm during 5 minutes with stretching.

The intervention in the VF group, the frequency of training will be 3 sessions per week on alternate days, the training will consist of 20 minutes of warm up, then the prinicpal work Aerobic training: 20 minutes of treadmill walking will be performed. Strength training with VF (20-25 min) as recommended by Chow et al.

1. Aerobic training: 20 minutes of treadmill walking will be performed. We will progress from 5-10 minutes until we reach a tolerable 20 minutes. The intensity will increase progressively until reaching 12-14 on the Borg scale.
2. Strength training with VF (20-25 min) following the recommendations of Chow et al (74):

i.Sets: start with 1 set to consolidate the technique, and progress to 3 sets. ii.Repetitions: start with 10-15 repetitions (at lower intensity) and progress to 8-12 repetitions.

iii.Intensity: start with a lower intensity (even 20-30%1RM) and progress to 70-80%1RM.

iv.Rest: Breaks between sets of 3-5 minutes should be taken to avoid muscle fatigue.

v.Exercises: Leg press on machine Balance and coordination training: 5-10 minutes. Throughout the training, focal vibration will be added with the V-Plus machine (Wintecare S.A. Chiasso (Switzerland)) on the rectus anterior, vastus medialis and vastus lateralis muscles with an intensity of 120 Hz and an amplitude of 1.2 mm finally return to calm during 5 minutes with stretching.

The intervention in the BFR group the frequency of training will be 3 sessions per week on alternate days, the training will consist of 20 minutes of warm up, then the strenght training with BFR 20-25 minutes with i. Series: start with 1 series to consolidate the technique, and progress to 3 series.

ii.Repetitions: a first series of 30 repetitions and 2 series of 15 repetitions.

iii.Intensity: the exercises will be performed at an intensity of 20%1RM and may reach 30%1RM if the subject can tolerate it.

iv.Rest: Breaks of 1 minute between sets. v.Exercises: Leg press on machine vi.Cuff occlusion pressure shall be set at 50% throughout the strength training portion of the workout.

vii.The cuff shall be placed on both lower extremities, inguinal. Balance and coordination training: 5-10 minutes, finally return to calm during 5 minutes with stretching.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary persons between 65 and 95 years of age.
* Have a walking speed ≤0.8 metres per second as this is characteristic of patients with or with onset of sarcopenia.
* Have a grip strength <30 kg for men and <20 kg for women as being characteristic of patients with or with onset of sarcopenia.

Exclusion Criteria:

* Severe untreated osteoporosis.
* Having suffered a bone fracture in the last year.
* Having had juvenile osteoporosis during adolescence or young adulthood.
* Active chronic pathology
* Uncontrolled arterial hypertension.
* Uncontrolled orthostatic hypotension.
* Severe acute respiratory failure.
* Diabetes mellitus with acute decompensation or uncontrolled hypoglycaemia.
* Endocrine, haematological and other associated rheumatic diseases.
* Mental health problems (schizophrenia, dementia, depression, etc.) or not being in full mental capacity.
* Patients with pharmacological treatments of glucocorticoids, anticoagulants and/or diuretics.
* Patients with coagulation problems or previous cardiac pathology.
* People with a body mass index (BMI) of 30 or more.
* Subjects with a systemic disease or any other pathology in which therapeutic exercise may be contraindicated.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical markers (BLOOD TESTS) | Change between baseline and post intervention
  Apelin, myostatin, IL6, plasma proteins, uric acid and creatinine.

SECONDARY OUTCOMES:
Physical Activity (PASE scale) | Change between baseline and post intervention
  Level of physical activity. This is a questionnaire administered by the researcher and answered by the participant (it can also be self-administered by the patient) where the level of physical activity in the participant's daily life is assessed.
Neuromuscular Function,Tensiomyography (Shrinkage time (Tc), and Radial displacement (Dm). | Change between baseline and post intervention
  Tensiomyography is an instrument which, at a given power, generates an involuntary muscle contraction in the muscle under examination. The contraction causes a movement of the muscle belly in a radial direction which is detected by a mechanical sensor placed just in contact with the muscle. The mechanical sensor collects the variables of contraction time (Tc) and radial displacement (Dm).
Neuromuscular Function, Myotonometry (Stiffness) | Change between baseline and post intervention
  Myotonometry is an instrument that assesses the viscoelasticity of tissue by means of a mechanical impulse in the muscle belly. The device generates a small mechanical impulse in the muscle belly and, depending on the response of the muscle belly to this stimulus, provides the variable stiffness.
Neuromuscular Function, Surface electromyography: (% RMS) | Change between baseline and post intervention
  Surface electromyography records the electrical activity that reaches the muscle in response to a nerve stimulus. The electrical activity of the above-mentioned muscles shall be collected during functional tests.
Neuromuscular Function, Manual Dinamometry. Pick force (kg) | Change between baseline and post intervention
  A hand-held dynamometer shall be used to assess the maximal force during an isometric contraction in the above movements. The participant shall exert force in the direction of movement and shall be resisted by the hand-held dynamometer to prevent movement and thus cause a maximal isometric contraction.
Neuromuscular Function, Handgrip (Kg) | Change between baseline and post intervention
  A hand-held dynamometer shall be used to assess the maximum grip force for 5 seconds. The participant shall squeeze the dynamometer as hard as possible and the dynamometer shall record the force applied.
Neuromuscular Function, Stabilometry | Change between baseline and post intervention
  This is a force platform that assesses balance in a standing position for 60 seconds while looking at a fixed point.
Neuromuscular Function, Ultrasound | Change between baseline and post intervention
  Ultrasound has been shown to be a valid and reliable tool for measuring cross-section in older people as well as an indicator of good health and reduced mortality. Ultrasound scans will be performed on a cross section at the level of the middle third of the muscle belly of the rectus femoris, vastus lateralis and vastus medialis muscles. The cross-sectional height, length and area of each image will be measured. Three images per muscle shall be taken and the mean of each image shall be obtained.
Fragility and independence (Barthel index) | Change between baseline and post intervention
  This is a questionnaire administered by the researcher and answered by the participant (it can also be self-administered by the patient) which assesses the participant's dependence on activities of daily living.
Fragility and independence (FRAIL scale) | Change between baseline and post intervention
  This is a questionnaire administered by the researcher and answered by the participant (it can also be self-administered by the patient) which assesses the participant's frailty in activities of daily living.
Fragility and independence (Falls Efficacy Scale I) | Change between baseline and post intervention
  This is a questionnaire administered by the researcher and answered by the participant (it can also be self-administered by the patient) where the fear of falling in activities of daily living is assessed.
Fragility and independence (SARC-F) | Change between baseline and post intervention
  It is a questionnaire administered by the researcher and answered by the participant (it can also be self-administered by the patient) that assesses muscle strength through an evaluation and scoring system in which patients record their ability in 5 parameters: strength, ability to walk, stand up from a chair, climb stairs and frequency of falls.
Functionality (Short Physical Performance Battery) | Change between baseline and post intervention
  It consists of a battery of three exercises with a maximum score of 4 points each. The first exercise assesses the participant's balance, the second exercise assesses walking speed and the third exercise assesses the strength of the lower limbs to stand up and sit down from the chair. The maximum SPPB score is 12 points indicating excellent functionality.
Functionality (Running speed in 4 metres) | Change between baseline and post intervention
  The participant's speed in covering 4 metres at their usual walking speed is assessed. The shorter the time, the faster the walking speed and therefore the better the functionality.
Functionality (Timed get up and go) | Change between baseline and post intervention
  The time it takes the participant to get up from a chair, walk 3 metres, turn around an obstacle (a cone) and sit back down in the chair is assessed. The less time the participant takes to perform the test, the better the functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain